CLINICAL TRIAL: NCT01960504
Title: BIOTRONIK - Safety and Clinical PerFormance of the Drug Eluting Absorbable Metal Scaffold (DREAMS 2nd Generation) in the Treatment of Subjects With de NOvo Lesions in NatiVE Coronary Arteries: BIOSOLVE-II
Brief Title: First in Man Study of the DREAMS 2nd Generation Drug Eluting Absorbable Metal Scaffold (BIOSOLVE-II)
Acronym: BIOSOLVE-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1209
Record Dates: First submitted 2013-10-06; First posted 2013-10-10 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis
Keywords: DREAMS; Drug Eluting Absorbable Metal Scaffold; Scaffold; Coronary Artery Disease; Myocardial Ischemia; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Myocardial Ischemia; Atherosclerosis | interventions — Percutaneous Coronary Intervention; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug Eluting Absorbable Metal Scaffold (Experimental): DREAMS 2nd Generation Drug Eluting Absorbable Metal Scaffold
  Interventions: Device: Percutaneous Coronary Intervention (DREAMS) stenting

INTERVENTIONS:
Device: Percutaneous Coronary Intervention (DREAMS) stenting
  Other Names: DREAMS 2nd Generation Drug Eluting Absorbable Metal Scaffold

SUMMARY:
BIOSOLVE-II is a prospective, international, multicenter, First in Man study. The purpose of this study is to assess the safety and clinical performance of the drug eluting absorbable metal scaffold (DREAMS 2nd Generation).

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years and < 80 years of age
* Written subject informed consent available prior to PCI
* Subjects with stable or unstable angina pectoris or documented silent ischemia
* Subject eligible for PCI
* Subject acceptable candidate for coronary artery bypass surgery
* Subjects with a maximum of two single lesions in two separate coronary arteries which have to be de novo lesions.
* Reference vessel diameter between 2.2-3.8 mm by visual estimation
* Target lesion length ≤ 21 mm by visual estimation
* Target lesion stenosis by visual estimation, assisted by QCA / IVUS: > 50% - < 100%
* Eligible for Dual Anti Platelet Therapy (DAPT)

Exclusion Criteria:

* Pregnant or breast-feeding females or females who intend to become pregnant during the time of the study
* Evidence of myocardial infarction within 72 hours prior to index procedure
* Subjects with a ≥2 fold CK level or in absence of CK a ≥3 fold CKMB level above the upper range limit within 24 hours prior to the procedure
* Unprotected left main coronary artery disease
* Three-vessel coronary artery disease at time of procedure
* Thrombus in target vessel
* Subject is currently participating in another study with an investigational device or an investigational drug and has not reached the primary endpoint yet
* Planned interventional treatment of any non-target vessel within 30 days post-procedure
* Subjects on dialysis
* Planned intervention of the target vessel within 6-month after the index procedure
* Ostial target lesion (within 5.0 mm of vessel origin)
* Target lesion involves a side branch >2.0 mm in diameter
* Documented left ventricular ejection fraction (LVEF) ≤ 30%
* Heavily calcified lesion
* Target lesion is located in or supplied by an arterial or venous bypass graft
* The target lesion requires treatment with a device other than the pre-dilatation balloon prior to scaffold placement (including but not limited to, rotational atherectomy, cutting balloon etc.)
* Known allergies to: Acetylsalicylic Acid (ASA), Heparin, Contrast medium, Sirolimus, or similar drugs; or the scaffold material
* Impaired renal function (serum creatinine > 2.5 mg/dl or 221 mmol/l, determined within 72 hours prior to intervention)
* Subject is receiving oral or intravenous immuno-suppressive therapy (e.g., inhaled steroids are not excluded) or has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, but not including diabetes mellitus)
* Proximal or distal to the target lesion located stenosis that might require future revascularization or impede run off detected during diagnostic angiography
* Life expectancy less than 1 year
* Planned surgery or dental surgical procedure within 6 months after index procedure
* In the investigators opinion subjects will not be able to comply with the follow-up requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
In segment Late Lumen Loss | 6 months post index procedure

SECONDARY OUTCOMES:
Target Lesion Failure (TLF), defined as composite of cardiac death, target vessel Q-wave or non-Q-wave Myocardial Infarction (MI), Coronary Artery Bypass Graft (CABG), clinically driven Target Lesion Revascularisation (TLR) | 1, 6, 12, 24 and 36 months
Scaffold thrombosis rate | 1, 6, 12, 24 and 36 months
In-scaffold and in-segment Binary Restenosis Rate | 6 and 12 months
In-scaffold and in-segment Percent Diameter Stenosis | 6 and 12 months
Late Lumen Loss in segment | 12 months
Late Lumen Loss in scaffold | 6 and 12 months
Procedure success | During the hospital stay to a maximum of the first seven days post index procedure
  Procedure Success defined as achievement of a final diameter stenosis of <30% by QCA, using any percutaneous method, without the occurrence of death, Q-wave or WHO defined non-Q-wave, or repeat revascularization of the target lesion during the hospital stay.
Device success | Day 0
  Device Success is defined as a final residual diameter stenosis of <30% by QCA, using the assigned device only
  * successful delivery of the scaffold to the target lesion site in the coronary artery
  * appropriate scaffold deployment
  * successful removal of the device
  * safe removal of the device in case of deployment failure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haude, MD, Principal Investigator — Städtische Kliniken Neuss
Locations (13):
- OLV-Ziekenhuis Aalst, Aalst, Belgium
- Brazil (2):
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Instituto do Coração - HCFMUSP, São Paulo
- Aarhus University Hospital, Aarhus, Denmark
- Germany (4):
  - Universitäts-Herzzentrum Freiburg Bad Krozingen, Bad Krozingen
  - Segeberg Kliniken GmbH, Herzzentrum, Bad Segeberg
  - Vivantes Klinikum, Berlin
  - Städtische Kliniken Neuss - Lukaskrankenhaus, Neuss
- Thoraxcentrum Twente, Enschede, Netherlands
- National Heart Centre Singapore, Mistri Wing, Singapore
- Hospital Clinico San Carlos, Madrid, Spain
- Switzerland (2):
  - University Hospital Basel, Basel
  - CHUV - Centre Hospitalier Universitaire Vaudois, Lausanne

REFERENCES:
- [Derived] Ozaki Y, Kuku KO, Sakellarios A, Haude M, Hideo-Kajita A, Desale S, Siogkas P, Sioros S, Ince H, Abizaid A, Tolg R, Lemos PA, von Birgelen C, Christiansen EH, Wijns W, Escaned J, Michalis L, Fotiadis DI, Djikstra J, Waksman R, Garcia-Garcia HM. Impact of Endothelial Shear Stress on Absorption Process of Resorbable Magnesium Scaffold: A BIOSOLVE-II Substudy. Cardiovasc Revasc Med. 2021 Aug;29:9-15. doi: 10.1016/j.carrev.2021.04.003. Epub 2021 Apr 9. PMID 33863661
- [Derived] Ueki Y, Raber L, Otsuka T, Rai H, Losdat S, Windecker S, Garcia-Garcia HM, Landmesser U, Koolen J, Byrne R, Haude M, Joner M. Mechanism of Drug-Eluting Absorbable Metal Scaffold Restenosis: A Serial Optical Coherence Tomography Study. Circ Cardiovasc Interv. 2020 Mar;13(3):e008657. doi: 10.1161/CIRCINTERVENTIONS.119.008657. Epub 2020 Feb 25. PMID 32093514
- [Derived] Ozaki Y, Garcia-Garcia HM, Hideo-Kajita A, Kuku KO, Haude M, Ince H, Abizaid A, Tolg R, Lemos PA, von Birgelen C, Christiansen EH, Wijns W, Escaned J, Waksman R. Serial 3-Dimensional Optical Coherence Tomography Assessment of Jailed Side-Branch by Second-Generation Drug-Eluting Absorbable Metal Scaffold (from the BIOSOLVE-II Trial). Am J Cardiol. 2019 Apr 1;123(7):1044-1051. doi: 10.1016/j.amjcard.2018.12.029. Epub 2019 Jan 4. PMID 30683424
- [Derived] Garcia-Garcia HM, Haude M, Kuku K, Hideo-Kajita A, Ince H, Abizaid A, Tolg R, Lemos PA, von Birgelen C, Christiansen EH, Wijns W, Escaned J, Dijkstra J, Waksman R. In vivo serial invasive imaging of the second-generation drug-eluting absorbable metal scaffold (Magmaris - DREAMS 2G) in de novo coronary lesions: Insights from the BIOSOLVE-II First-In-Man Trial. Int J Cardiol. 2018 Mar 15;255:22-28. doi: 10.1016/j.ijcard.2017.12.053. Epub 2017 Dec 28. PMID 29292064
- [Derived] Haude M, Ince H, Abizaid A, Toelg R, Lemos PA, von Birgelen C, Christiansen EH, Wijns W, Neumann FJ, Kaiser C, Eeckhout E, Lim ST, Escaned J, Onuma Y, Garcia-Garcia HM, Waksman R. Sustained safety and performance of the second-generation drug-eluting absorbable metal scaffold in patients with de novo coronary lesions: 12-month clinical results and angiographic findings of the BIOSOLVE-II first-in-man trial. Eur Heart J. 2016 Sep 14;37(35):2701-9. doi: 10.1093/eurheartj/ehw196. Epub 2016 May 17. PMID 27190094
- [Derived] Haude M, Ince H, Abizaid A, Toelg R, Lemos PA, von Birgelen C, Christiansen EH, Wijns W, Neumann FJ, Kaiser C, Eeckhout E, Lim ST, Escaned J, Garcia-Garcia HM, Waksman R. Safety and performance of the second-generation drug-eluting absorbable metal scaffold in patients with de-novo coronary artery lesions (BIOSOLVE-II): 6 month results of a prospective, multicentre, non-randomised, first-in-man trial. Lancet. 2016 Jan 2;387(10013):31-9. doi: 10.1016/S0140-6736(15)00447-X. Epub 2015 Oct 12. PMID 26470647